CLINICAL TRIAL: NCT06317311
Title: A Phase 2, Multicenter, Open-label, Single Arm Study of Dostarlimab Plus Carboplatin-paclitaxel Followed by Dostarlimab Monotherapy in Japanese Patients With Primary Advanced or Recurrent Endometrial Cancer (RUBY-J)
Brief Title: A Study of Dostarlimab in Combination With Carboplatin-paclitaxel in Japanese Participants With Primary Advanced or Recurrent Endometrial Cancer
Acronym: RUBY-J
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 221968
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma
Keywords: Endometrial cancer; Dostarlimab; Carboplatin; Paclitaxel
MeSH Terms: conditions — Carcinoma; Endometrial Neoplasms | interventions — dostarlimab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dostarlimab- Carboplatin-Paclitaxel followed by Dostarlimab Monotherapy (Experimental)
  Interventions: Biological: Dostarlimab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Dostarlimab — Dostarlimab is administered via intravenous (IV) infusion at a dose of 500 milligram (mg) for first 6 cycles (each cycle is of 21 days) followed by 1,000 mg from cycle 7 (each cycle is of 42 days)
Drug: Carboplatin — Carboplatin is administered IV at a dose of Area under the concentration time curve (AUC) 5 milligram*millilitre/ minute (mg•mL/min) for cycles 1 to 6 (each cycle is of 21 days)
Drug: Paclitaxel — Paclitaxel is administered IV at a dose of 175 milligram per meter square (mg/m2) for cycles 1 to 6 (each cycle is of 21 days)

SUMMARY:
The goal of this clinical trial is to understand the effectiveness of dostarlimab and carboplatin-paclitaxel followed by dostarlimab monotherapy in participants with endometrial cancer

ELIGIBILITY:
Inclusion Criteria:

1. Participant has histologically or cytologically proven endometrial cancer with recurrent or advanced disease.
2. Participant has molecular subtype of defective mismatch repair/microsatellite instability high (dMMR/MSI-H) or mismatch repair proficient/microsatellite stable (MMRp/MSS) determined.
3. Participant must have primary Stage III or Stage IV disease or first recurrent endometrial cancer with a low potential for cure by radiation therapy or surgery alone or in combination, and presence of at least one measurable lesion per RECIST 1.1 based on Investigator's assessment.
4. Participant is not pregnant or breastfeeding and agrees to use a highly effective contraceptive method during the study period if a woman of childbearing potential (WOCBP).
5. Participant has an Eastern Cooperative Oncology Group Performance status (ECOG PS) of 0 or 1.
6. Participant has adequate organ function, as assessed by hematologic, renal, hepatic and coagulation parameters.

Exclusion Criteria:

1. Participant has a concomitant malignancy, or participant has a prior non-endometrial invasive malignancy who has been disease-free for <3 years or who received any active treatment in the last 3 years for that malignancy. Non-melanoma skin cancer is allowed.
2. Participant has any medical history of interstitial lung disease or pneumonitis.
3. Participant has cirrhosis or current unstable liver or biliary disease.
4. Participant has known uncontrolled central nervous system metastases, carcinomatosis meningitis, or both.
5. Participant has a diagnosis of immunodeficiency.
6. Participant has received prior therapy with an anti- Programmed death protein 1 (PD-1), anti- Programmed death ligand 1 (PD-L1), anti- Programmed death ligand 2 (PD-L2), or anti- Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) agent.
7. Participant has not recovered adequately from AEs.
8. Participant has received prior anticancer therapy (chemotherapy, targeted therapies, hormonal therapy, radiotherapy, or immunotherapy) within 21 days or <5 times the half-life of the most recent therapy prior to the first dose of study intervention, whichever is shorter.
9. Participant has received any live vaccine within 30 days of the first dose of study intervention. Vaccination against coronavirus disease 2019 (COVID-19) using vaccines that are authorized via the appropriate regulatory mechanisms are not exclusionary.
10. Participant has HBsAg positive, or HCV RNA positive.
11. Participant is known HIV infection.
12. Participant is currently participating and receiving study intervention or has participated in a study of an investigational agent and received study intervention or used an investigational device within 4 weeks of the first dose of treatment.
13. Participant with contraindication to carboplatin and paclitaxel.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 41 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Durable response rate for 12 months (DRR12) assessed by Blinded independent central review (BICR) | Approximately 18 months
  DRR12 is defined as the proportion of participants with Complete Response (CR) or Partial Response (PR) lasting greater than or equal to (≥) 12 months, per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
DRR12 per RECIST 1.1, assessed by investigator | Approximately 18 months
Progression-free survival (PFS) per RECIST 1.1, assessed by BICR and investigator | Up to approximately 3 years
  PFS is defined as the time from the date of first dose to the earlier date of assessment of progression or death by any cause
Overall survival (OS) | Up to approximately 3 years
  OS is defined as time from first dose of study intervention to death from any cause
Overall response rate (ORR) per RECIST 1.1 assessed by BICR | Up to approximately 3 years
  ORR is achieving a best overall response (BOR) of CR or PR. BOR is defined as the best confirmed response [CR > PR > Stable disease (SD) > Progressive Disease (PD) > Not evaluable (NE)] from treatment start date until disease progression, death or initiation of next line of therapy, whichever is earlier
ORR per RECIST 1.1 assessed by investigator | Up to approximately 3 years
Disease control rate (DCR) per RECIST 1.1 assessed by BICR | Up to approximately 3 years
  Achieving a BOR of CR, PR, or SD, defined as the best confirmed response (CR > PR > SD) from treatment start date until disease progression, death or initiation of next line of therapy, whichever is earlier
DCR per RECIST 1.1 assessed by investigator | Up to approximately 3 years
Duration of response (DOR) per RECIST 1.1 assessed by BICR | Up to approximately 3 years
  DOR is defined as the time from the date of first documented objective response to the date of first documented PD or death, whichever comes first
DOR per RECIST 1.1 assessed by investigator | Up to approximately 3 years
Maximum concentration (Cmax) for dostarlimab | Up to 67 weeks
Minimum concentration (Cmin) for dostarlimab | Up to 67 weeks
Number of participants with adverse events (AEs), Immune-related adverse events (irAEs), and serious adverse events (SAEs) by severity | Up to approximately 3 years
Number of participants AEs, irAEs, and SAEs leading to dose modifications such as dose delay or study intervention discontinuation | Up to approximately 3 years
Number of participants with AEs leading to death | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Locations (16):
- Japan (16):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/